CLINICAL TRIAL: NCT05627245
Title: Phase 1/Expansion Study of Tazemetostat Plus Belinostat for the Treatment of Relapsed or Refractory Lymphoma
Brief Title: Testing the Safety of the Anti-cancer Drugs Tazemetostat and Belinostat in Patients With Lymphomas That Have Resisted Treatment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-05327; NCI-2022-05327 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CUMC-AAAT9882; 10500 (Other: Yale University Cancer Center LAO); 10500 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2022-11-23; First posted 2022-11-25 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Recurrent Follicular Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Recurrent T-Cell Non-Hodgkin Lymphoma; Recurrent Transformed Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Refractory Follicular Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Refractory T-Cell Non-Hodgkin Lymphoma; Refractory Transformed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell | interventions — belinostat; Biopsy; Specimen Handling; Pharmacogenomic Variants; Magnetic Resonance Spectroscopy; tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (tazemetostat, belinostat) (Experimental): Patients receive tazemetostat PO BID on days 2-21 of cycle 1 and days 1-21 of subsequent cycles, and belinostat IV over 30-180 minutes on days 1-5 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Patients may undergo a tumor biopsy during screening and on study (dose-expansion only). Patients undergo blood sample collection while on study and CT or PET/CT scan throughout the study.
  Interventions: Drug: Belinostat; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Pharmacokinetic Study; Procedure: Positron Emission Tomography and Computed Tomography Scan; Drug: Tazemetostat

INTERVENTIONS:
Drug: Belinostat — Given IV
  Other Names: Beleodaq; PXD 101; PXD-101; PXD101
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Pharmacokinetic Study — Pharmacokinetic study
  Other Names: PHARMACOKINETIC; PK Study
Procedure: Positron Emission Tomography and Computed Tomography Scan — Undergo PET-CT
  Other Names: PET-CT Scan; PET/CT SCAN; Positron Emission Tomography/Computed Tomography
Drug: Tazemetostat — Given PO
  Other Names: E 7438; E-7438; E7438; EPZ 6438; EPZ-6438; EPZ6438

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of combination therapy with tazemetostat and belinostat in treating patients with lymphoma that has come back after a period of improvement (relapsed) or that does not respond to treatment (refractory). Tazemetostat is in a class of medications called EZH2 inhibitors. The EZH2 gene provides instructions for making a type of enzyme called histone methyltransferase which is involved in gene expression and cell division. Blocking EZH2 may help keep cancer cells from growing. Belinostat is in a class of medications called histone deacetylase inhibitors. Histone deacetylases are enzymes needed for cell division. Belinostat may kill cancer cells by blocking histone deacetylase. It may also prevent the growth of new blood vessels that tumors need to grow and may help make cancer cells easier to kill with other anticancer drugs. There is some evidence in animals and in living human cells that combination therapy with tazemetostat and belinostat can shrink or stabilize cancer, but it is not known whether this will happen in people. This trial may help doctors learn more about treatment of patients with relapsed or refractory lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) of tazemetostat and belinostat in combination in patients with relapsed or refractory lymphoma. (Phase I: Dose escalation) II. Evaluate the safety and toxicity of the combination tazemetostat and belinostat. (Phase I: Dose escalation) III. Assess the safety and tolerability of tazemetostat and belinostat in patients with germinal-center derived B-cell lymphoma (follicular lymphoma, transformed disease, diffuse large B-cell lymphoma germinal center B-cell type [GC-DLBCL] defined by Hans criteria), and T-cell lymphomas. (Phase I: Dose expansion) IV. Assess the impact of EZH2, CREBBP, and EP300 mutations on response to dual epigenetic targeting. (Phase I: Dose expansion)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To evaluate the pharmacokinetic profile for tazemetostat and belinostat when given as a combination.

III. Define the overall response rate (ORR), progression free survival (PFS), and duration of response (DOR) in patients with relapsed or refractory EZH2 mutated and EZH2 wild-type germinal-center derived B-cell lymphoma (follicular lymphoma, transformed disease, GC-DLBCL defined by Hans criteria), as well as T-cell lymphomas.

IV. To describe the maximum number of cycles received, the number of dose reductions and delays at the MTD.

EXPLORATORY OBJECTIVES:

I. Determine a biomarker for response by assessing the basal mutation and gene expression status of key epigenetic regulators and correlating this signature with the response to the combination.

II. Determine the change in gene expression in tumor tissue following exposure the combined epigenetic therapy.

III. Determine the effect of combination epigenetic therapy on modulation of acetylation and methylation of histone K27.

IV. Determine the effect of combination epigenetic therapy on modulation of the immune response.

OUTLINE: This is a phase I dose-escalation study of tazemetostat and belinostat followed by a dose-expansion study.

Patients receive tazemetostat orally (PO) twice daily (BID) on days 2-21 of cycle 1 and days 1-21 of subsequent cycles, and belinostat intravenously (IV) over 30-180 minutes on days 1-5 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients may undergo a tumor biopsy during screening and on study (dose-expansion only). Patients undergo blood sample collection while on study and computed tomography (CT) or positron emission tomography (PET)/CT scan throughout the study.

After completion of study treatment, patients are followed up at 4 weeks, then every 3 months for a year or until they begin a new treatment for their disease.

ELIGIBILITY:
Inclusion Criteria:

* DOSE ESCALATION PHASE: Patients with relapsed or refractory non-Hodgkin lymphoma including both B-cell non-Hodgkin lymphoma (NHL) and T-cell NHL. Refractory cutaneous T-cell lymphoma (CTCL) will be allowed if greater or equal to stage 1B and have previously failed two systemic therapies
* DOSE EXPANSION PHASE: Patients with relapsed or refractory follicular, transformed lymphoma or germinal center B-cell diffuse large B-cell Lymphoma (GCB-DLBCL) as defined by Hans criteria, as well as T-cell lymphomas. For patients with B-cell lymphomas, equal numbers of patients will be enrolled onto one of 2 arms: (1) mutated EZH2 or (2) wild-type EZH2. EZH2 mutations will be identified by polymerase chain reaction (PCR)
* Patients must not be eligible for, or have refused, stem cell transplantation or chimeric antigen receptor T-cell (CAR T-cell) therapy
* Patients who have undergone 1-5 prior treatments of any type (progression after transplant/cellular therapy allowed) are eligible
* Patients must have measurable disease according to the Lugano classification
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of tazemetostat in combination with belinostat in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,000/mcL

  * If there is documented lymphomatous involvement of the bone marrow as assessed by bone marrow biopsy within 90 days prior to registration, participants should have: absolute neutrophil count (ANC) >= 0.75 × 10^9/L
* Platelets >= 75,000/mcL

  * If there is documented lymphomatous involvement of the bone marrow as assessed by bone marrow biopsy within 90 days prior to registration, participants should have: platelets >= 50 x 10^9/L
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN); unless due to Gilbert's disease, hemolysis, or lymphomatous involvement of liver, in which case total bilirubin should be =< 5 x institutional ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN; unless due to Gilbert's disease, hemolysis, or lymphomatous involvement of liver, in which case AST(SGOT)/ALT(SGPT) should be =< 5 x institutional ULN
* Glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Patients whose lymphoma has transformed from a less aggressive histology remain eligible
* Patients should be New York Heart Association Functional Classification of class II or better
* Patients must have a QT interval corrected by Fridericia's formula (QTcF) =< 450 msec
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption, such as malabsorption syndrome or major resection of the stomach or bowels
* The effects of tazemetostat and belinostat on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use two reliable methods of contraception simultaneously prior to study entry and for the duration of study participation and for 6 months after the last dose of the study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of tazemetostat and belinostat administration. Male participants must not donate semen or sperm from first dose of study drug, during study treatment (including during dose interruptions), and for 3 months after study drug discontinuation
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* Patients that have received prior chemotherapy or radiotherapy must have completed their last treatment at least 2 weeks before entering the study. Rituximab given between EZH2 analysis and initiation of study drugs will be allowed

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients with active central nervous system (CNS) metastases, including lymphomatous meningitis, as the study drugs are not known to effectively treat CNS disease
* History of allergic reactions attributed to belinostat or tazemetostat, or to compounds of similar chemical or biologic composition to these agents
* Patients receiving any medications or substances that are strong or moderate inhibitors or inducers of CYP3A4 within 14 days prior to study treatment are ineligible. Patients receiving strong UGT1A1 inhibitors are ineligible due to expected increased exposure to belinostat and potential for increased toxicity. Because the list of these agents is constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with known UGT1A1 genetic polymorphisms, such as UGT1A1*28, are excluded as they can have reduced UGTA1A activity and may be at risk for increased belinostat exposure
* Patients with uncontrolled intercurrent illness
* Pregnant women are excluded from this study because belinostat, as an HDAC inhibitor, and tazemetostat, as an EZH2 inhibitor, both have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with belinostat and tazemetostat, breastfeeding should be discontinued if the mother is treated with belinostat and tazemetostat. Women of childbearing potential must have negative urine or serum pregnancy test to be eligible for this study
* Systemic steroids that have not been stabilized to the equivalent of =< 10 mg/day prednisone prior to the start of the study drugs and throughout the study. Patients are allowed to receive dexamethasone as premedication during belinostat infusion
* Has thrombocytopenia, neutropenia, or anemia of grade >= 3 (per Common Terminology Criteria for Adverse Events [CTCAE] 5.0 criteria) or any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS)
* Has abnormalities known to be associated with MDS (e.g. 5q deletion [del 5q], chromosome 7 abnormality [chr 7 abn]) and multiple primary neoplasms (MPN) (e.g. JAK2 V617F) observed in cytogenetic testing and deoxyribonucleic acid (DNA) sequencing
* Has a prior history of T lymphoblastic lymphoma/T acute lymphoblastic leukemia (T-LBL/T-ALL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (Dose escalation) | Up to end of cycle 1 (Cycles = 21 days)
  Defined as the highest dose level at which < 33% of the dose cohort (0 of 3 or 1 of 6) experience a dose-limiting toxicity in the first cycle.

SECONDARY OUTCOMES:
Disease response | Following cycle 2 and 6, and every 3-6 cycles, assessed up to 1 year after completion of study treatment
  Will be assessed by positron emission tomography/computed tomography scan following cycle 2 and 6, and then every 3-6 cycles. Response will be defined by the Lugano Classification.
Overall response rate | Up to 1 year after completion of study treatment
  Defined as complete response + partial response. Will be estimated and the exact 95% confidence interval will be constructed based on binomial distribution.
Progression-free survival | From time to enrollment to progression or death, assessed up to 1 year after completion of study treatment
  Will be estimated by the Kaplan-Meier method and compared by the log-rank test.
Overall survival | From time to enrollment to death, assessed up to 1 year after completion of study treatment
  Will be estimated by the Kaplan-Meier method and compared by the log-rank test.
Duration of response | From first response to relapse or death, assessed up to 1 year after completion of study treatment
  Will be estimated by the Kaplan-Meier method.
Total number of cycles | Up to 2 years
  The mean and range will be calculated.
Number of dose delays | Up to 2 years
  The mean and range will be calculated.
Number of dose reductions | Up to 2 years
  The mean and range will be calculated.
Pharmacokinetic profile for tazemetostat and belinostat | Cycle 1, day 1 (C1D1) (belinostat only) and C2D1
  Plasma concentrations of both tazemetostat and belinostat using area under the "concentration time" curve, maximum concentration, time to maximum concentration, and half-life will be calculated for the two study drugs.
Incidence of adverse events | Up to 4 weeks after completion of study treatment
  National Cancer Institute toxicity Grade 3 and Grade 4 laboratory abnormalities will be listed. Summary statistics will be provided for all laboratory values.

OTHER OUTCOMES:
Modulation in immune function | During cycle 1 (Cycles = 21 days)
  Will be presented in descriptive terms.
Histone acetylation and methylation | Up to 2 years
  Will be assessed separately for the wild type and the mutant groups and will be compared using a two-sample Wilcoxon rank-sum test.
Gene signature biomarker for response | Up to 2 years
  Will be evaluated next generation sequencing and presented in descriptive terms. Gene signature biomarker data analysis will be completed using Lasso-based elastic net method.
Modulation of histone acetylation and methylation | Up to 2 years
  Will be presented in descriptive terms.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Amengual, Principal Investigator — Yale University Cancer Center LAO
Locations (11):
- United States (11):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Yale University, New Haven, Connecticut
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm